CLINICAL TRIAL: NCT03002129
Title: FLuid Responsiveness Prediction Using EXtra Systoles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof.dr.T.W.L.Scheeren, prof.dr., University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLEx study
Record Dates: First submitted 2016-12-15; First posted 2016-12-23 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Bypass Graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fluid challenge (Other)
  Interventions: Other: fluid challenge

INTERVENTIONS:
Other: fluid challenge — At two pre-defined time points during the procedure, enrolled patients will receive a fluid bolus of 5 ml/kg during 5 minutes

SUMMARY:
In this study, the investigators propose to investigate a novel technique for fluid responsiveness prediction. It is based on the occurrence of an extra systole, which induces a preload variation: Extra systoles are comprised by, first, the premature/ectopic beat with decreased cardiac preload, then, the post-ectopic beat with moderately increased preload.

Consequently, the post ectopic beat is associated with a Frank-Starling curve right shift but is otherwise a normal sinus beat. As such, the post-ectopic beat elucidates and predicts the hemodynamic effect of increasing preload, i.e. giving fluids

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring elective CABG or OPCAB surgery
* Patient's age ≥ 18 years

Exclusion Criteria:

* Patient refusal
* Pregnancy
* EF < 35%
* End stage kidney failure (defined by the need for haemodialysis)
* Patients with atrial fibrillation or frequent and coupled extra systoles (e.g. trigemini)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
fluid challenge response in stroke volume | during operation
  To investigate if post-ectopic induced changes in blood pressure before a fluid bolus (5 ml/kg) predicts the fluid induced change in cardiac stroke volume

CONTACTS AND LOCATIONS:
Locations (1):
- Universitu Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holmgaard F, Vistisen ST, Ravn HB, Scheeren TWL. The response of a standardized fluid challenge during cardiac surgery on cerebral oxygen saturation measured with near-infrared spectroscopy. J Clin Monit Comput. 2020 Apr;34(2):245-251. doi: 10.1007/s10877-019-00324-w. Epub 2019 May 28. PMID 31134474
- [Derived] Vistisen ST, Berg JM, Boekel MF, Modestini M, Bergman R, Jainandunsing JS, Mariani MA, Scheeren TWL. Using extra systoles and the micro-fluid challenge to predict fluid responsiveness during cardiac surgery. J Clin Monit Comput. 2019 Oct;33(5):777-786. doi: 10.1007/s10877-018-0218-0. Epub 2018 Nov 9. PMID 30414054